CLINICAL TRIAL: NCT01006694
Title: Paraprofessional Treatment of Depression in Vietnam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vietnam Veterans of America Foundation (Other)
Collaborators: RAND (Other); Vanderbilt University (Other)
Responsible Party: Principal Investigator, Bahr Weiss, Associate Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20090928.1
Record Dates: First submitted 2009-11-02; First posted 2009-11-03 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Depressive Symptoms
Keywords: depression; collaborative care; Vietnam; behavioral activation
MeSH Terms: conditions — Depression | interventions — Dosage Forms; Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Guideline Antidepressant Medication (Active Comparator): Guideline Antidepressant Medication, following the VN National Mental Health plan.
  Interventions: Drug: Guideline Antidepressant Medication
- Behavioral Activation + Medication (Experimental): Psychoeducation, behavioral activation therapy, and medication delivered within a collaborative care model.
  Interventions: Other: Behavioral Activation + Medication

INTERVENTIONS:
Other: Behavioral Activation + Medication — Psychoeducation, behavioral activation therapy, and medication delivered within a collaborative care model.
  Other Names: BA + SSRI
  Arms: Behavioral Activation + Medication
Drug: Guideline Antidepressant Medication — Guideline Antidepressant Medication, following the VN National Mental Health plan.
  Arms: Guideline Antidepressant Medication

SUMMARY:
Trained para-professional health care workers will implement a stepped-care model of depression care in commune health stations in Vietnam.

DETAILED DESCRIPTION:
This project focuses on evaluation of a collaborative care system for treatment of depression in Vietnam. This system involves training para-professional health care workers in a stepped-care model system of depression care to be implemented in commune health stations in Vietnam.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=18
2. Depression Diagnosis

Exclusion Criteria: active psychosis, mania, substance abuse, suicidal behaviors, cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 473 (Actual)
Dates: Start 2010-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Change across time (random effects slope) in depressive symptoms, as assessed by the PHQ-9 questionnaire | 0, 6, 12, 24 weeks
  The PHQ-9 (Patient Health Questionnaire-9) assesses depressive symptoms, over the last two weeks. It is assessed at 0, 6, 12, 24 weeks. The outcome target is the linear and quadratic change slopes across these 4 time points.

SECONDARY OUTCOMES:
Change across time (random effects slope) in anxiety symptoms, as assessed by the GAD-7 questionnaire | 0, 6, 12, 24 weeks
  The GAD-7 (General Anxiety Disorder-7) assesses anxiety symptoms, over the last two weeks. It is assessed at 0, 6, 12, 24 weeks. The outcome target is the linear and quadratic change slopes across these 4 time points.
Change across time (random effects slope) in physical health, as assessed by the SF-12 questionnaire, Physical Health subscale | 0, 6, 12, 24 weeks
  The SF-12 questionnaire, Physical Health subscale, assesses physical health functioning. It is assessed at 0, 6, 12, 24 weeks. The outcome target is the linear and quadratic change slopes across these 4 time points.
Change across time (random effects slope) in mental health, as assessed by the SF-12 questionnaire, Mental Health subscale | 0, 6, 12, 24 weeks
  The SF-12 questionnaire, Mental Health subscale, assesses mental health functioning. It is assessed at 0, 6, 12, 24 weeks. The outcome target is the linear and quadratic change slopes across these 4 time points.
Change across time (random effects slope) in behavioral activation skills and behaviors, as assessed by the BADS questionnaire. | 0, 6, 12, 24 weeks
  The BADS (Behavioral Activation for Depression Scale) questionnaire assesses behavioral activation-related skills and behaviors. It is assessed at 0, 6, 12, 24 weeks. The outcome target is the linear and quadratic change slopes across these 4 time points.
"Substantial improvement" in depressive symptoms, as assessed by the PHQ-9 | 6, 12, 24 weeks
  Rates of substantial symptomatic improvement (50% or greater reduction in PHQ-9 scores from baseline), to (a) 6 weeks, (b) 12 weeks, (c) 24 weeks.
"Depression remission", as assessed by the PHQ-9 | 6, 12, 24 weeks
  Depression remission (PHQ-9<5), at (a) 6 weeks, (b) 12 weeks, (c) 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: victoria ngo, phd, Principal Investigator — RAND
Locations (2):
- Vietnam (2):
  - Khanh Hoa Provincial Hospital, Nha Trang, Khanh Hoa
  - Danang Psychiatric Hospital, Da Nang